CLINICAL TRIAL: NCT03193359
Title: A Multicenter, Open-label, Safety, Tolerability and Efficacy Study of BOTOX® (Botulinum Toxin Type A) as Headache Prophylaxis in Chinese Patients With Chronic Migraine
Brief Title: Open Label Study of BOTOX® (Botulinum Toxin Type A) as Headache Prophylaxis in Chinese Patients With Chronic Migraine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Corporate Decision
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1313-302-008
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BOTOX® (Experimental): BOTOX® (botulinum toxin Type A) 155U to 195U intramuscular (IM) injections to head/neck areas at Day 0 and Week 12.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A (BOTOX®) IM 155U to 195U injections in head/neck areas.
  Other Names: BOTOX®; onabotulinumtoxinA

SUMMARY:
This study is an open-label extension study to evaluate the safety, tolerability and efficacy of BOTOX® as headache prophylaxis in Chinese patients with chronic migraine who have successfully completed the double-blind study: 1313-301-008.

ELIGIBILITY:
Inclusion Criteria:

-Has successfully completed the double-blind study (1313-301-008).

Exclusion Criteria:

* Has met any of the withdrawal criteria in the double-blind study or has clinical significant abnormal laboratory or electrocardiogram (ECG) findings
* Headache attributable to another disorder (eg, cervical dystonia, craniotomy, head/neck trauma)
* Any medical condition that may put the patient at increased risk with exposure to Botulinum Toxin Type A, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2021-09-09 (Estimated); Study Completion 2021-09-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | 24 Weeks
  An AE is any untoward medical occurrence in a patient or a participant using an investigational drug, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Percentage of Participants with AEs Leading to Discontinuation | 24 Weeks
Change from Baseline in Vital Signs | Baseline, Week 24
  Vital signs include blood pressure and pulse.
Change from Baseline in 12-Lead Electrocardiograms (ECGs) Parameters | Baseline, Week 24
  A standard 12-lead ECG will be performed at Baseline and Week 24.
Change from Baseline in Clinical Laboratory Parameters | Baseline, Week 24
  Blood samples will be collected at Baseline and Week 24 for standard clinical laboratory testing including hematology, chemistry, urinalysis an immunogenicity parameters.

SECONDARY OUTCOMES:
Change from Baseline in the Frequency of Headache Days during 28-Day Period Ending with Weeks 12 and 24 | Baseline, Weeks 12 and 24
  Mean change from Baseline (28-days prior to first treatment) in frequency (number) of headache days during the 28-day period ending with Weeks 12 and 24. A headache day was defined as a calendar day [00:00 to 23:59] for which the participant reported ≥ 4 continuous hours of headache per patient diary.
Change from Baseline in Total Cumulative Hours of Headache Days during 28-Day period | Baseline, Weeks 12 and 24
  Mean change from Baseline (28-days prior to first treatment) in the total cumulative hours of headache days during the 28-day period ending with Weeks 12 and 24. A headache day is defined as a day (00:00 to 23:59) with 4 or more continuous hours of headache per patient diary.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Lum, Study Director — Allergan

REFERENCES:
- See also: More Information — http://allerganclinicaltrials.com